CLINICAL TRIAL: NCT03294447
Title: The Association Between Fear of Falling and Fall Prevention Interventions Offered by an Occupational Therapist in a Geriatric Primary Care Setting
Brief Title: An Occupational Therapist Fall Prevention Intervention in a Geriatric Primary Care Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Western Michigan University (Other)
Responsible Party: Principal Investigator, Lydia Royeen, Senior Occupational Therapist, Rush University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15082105-IRB01
Record Dates: First submitted 2017-05-23; First posted 2017-09-27 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Fall Accident; Fall, Accidental
Keywords: Fear of falling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fall Prevention Intervention by OT (Experimental): Fall prevention interventions implemented by an OT in a geriatric primary care setting for a client immediately following the provider visit within the office.
  Interventions: Behavioral: Fall Prevention by the Occupational Therapist

INTERVENTIONS:
Behavioral: Fall Prevention by the Occupational Therapist — The interventions included education on adaptive equipment for household activities, adaptive equipment for activities of daily living, proper footwear in all environments, proper body mechanics, position changes, home environment set up, high fall risk activities, safety awareness, low vision and home exercises programs. In addition, discussion and education occurred to improve participation in valued occupations.

SUMMARY:
Purpose of the study: To identify if an intervention focused on decreasing fear of falling (FOF) in a geriatric primary care setting implemented by an occupational therapist (OT) has the potential to decrease falls and improve physical, psychological and social factors related to FOF.

The primary research question: Is there an association between fear of falling among geriatric populations and fall prevention interventions that are offered by occupational therapist in a geriatric primary care setting?

ELIGIBILITY:
Inclusion Criteria:

* cognitively intact with a score of 29/30 or higher on the Orientation Log (standardized assessment tool)
* living in the community
* English speaking
* had a fall or near fall in the past year

Exclusion Criteria:

* received OT services within the past 2 months

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
The Change of Falls Efficacy Scale-International (FES-I), standardized measure for fear of falling | One Time visit: 30-50 minutes
  The outcome measure is the change between the pre FES-I and post FES-I

CONTACTS AND LOCATIONS:
Overall Officials: Lydia Royeen, Masters, Principal Investigator — Rush University Medical Center
Locations (1):
- Geriatric Primary Care Clinic, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided